CLINICAL TRIAL: NCT01642862
Title: A Phase I, Randomized, Open Label, Mono-centered, Prospective Study to Evaluate the Pharmacokinetics of Different Formulations and Doses of Simvastatin in Healthy Subjects and in Subjects With Celiac Disease in Remission
Brief Title: Study for Identifying Optimal Simvastatin Formulation for Uniform Time to Maximum Plasma Concentration
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: University of Zurich (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CYPCEL-1103
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liquid formulation of Simvastatin (Experimental)
  Interventions: Drug: Simvastatin
- Tablet formulation of Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Comparison of pharmacokinetic parameters of different formulations (liquid vs tablet) and doses (20 or 40 mg) of simvastatin after single oral administration of the drug

SUMMARY:
The inter- and intra-variability in the pharmacokinetic parameters of different formulations and doses of simvastatin in healthy subjects and in subjects with celiac disease in remission will be evaluated. Additionally, baseline values of pharmacokinetic parameters of simvastatin for both study groups will be determined.

ELIGIBILITY:
Inclusion criteria:

* If the subject is female, she is eligible to enter and participate in this study if she is physiologically incapable of becoming pregnant or has a negative urine pregnancy test at screening and at baseline visit
* Negative Serology for Hepatitis B/C, HIV
* Non-OATP1B1*5 carriers
* Negative Serology for anti-transglutaminase IgA antibody, and normal levels of total IgA
* For subjects with celiac disease, also

  * Diagnosis of celiac disease confirmed by medical history, histological evaluation of small intestinal mucosa on small bowel biopsy, and abnormal anti-transglutaminase antibody titers
  * Followed a gluten-free diet for at least one year, as verified by normal anti-transglutaminase antibody levels, Marsh 0-1 score on a follow-up biopsy within the past 12 months, and absence of any clinical signs or symptoms of celiac disease observed at diagnosis

Exclusion criteria:

* Current smoker or quit smoking less than 2 years ago
* Female breastfeeding or disagrees to use an effective mechanical contraceptive method (e.g. diaphragm or nonhormonal intrauterine device in combination with preservative)
* Presence of any known on-going disease which is judged to be relevant according to the investigator, besides celiac disease for the cohort of celiac patients in remission
* State after operations of the stomach or bowel (exception: appendectomy)
* Participation in any other clinical trial with investigational or approved drugs within the last month before the study
* Regular alcohol consumption of more than 25 g / day
* Use of any prescription or non-prescription drugs (including herbal supplements) must be discontinued 30 days prior to study (exceptions: paracetamol and NSAIDs, not taken longer than 2 days in a row and not taken within the last 3 days before the study)
* Consumption of grapefruit, star fruit, grapefruit juice, or star fruit juice must be discontinued 7 days prior to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of simvastatin | 0, 15, 30, 60, 90, 120, 180 minutes post-dose
  Determination of time-dependent concentrations of simvastatin in collected serum of each subject following oral administration of two different formulations and two different doses of simvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Rogler, Prof MD PhD, Principal Investigator — University Hospital Zurich, Gastroenterology and Hepatology
Locations (1):
- University Hospital Zurich, University Hospital Zurich, Gastroenterology and Hepatology, Zurich, Canton of Zurich, Switzerland